CLINICAL TRIAL: NCT01840293
Title: Breast Cancer Proteomics and Molecular Heterogeneity
Status: Recruiting | Type: Observational
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Other Study IDs: ICORG 09-07
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Primary Breast Cancer; Recurrent/Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Primary Breast Cancer
- Recurrent/Metastatic Breast Cancer

SUMMARY:
Primary objective:

The primary objective is to define the proteomic and molecular characteristics of primary and recurrent/ metastatic breast tumours with special focus on the expression of S100 protein and the estrogen receptor (ER), progesterone receptor (PR) and epidermal growth factor receptor 2 (HER2) genes

Secondary objective:

* To expand our understanding of the complex molecular pathways dictating the progression of breast cancer and their response to different treatment regimes.
* To relate proteomic findings to survival data
* To identify potential serum markers of breast cancer progression

DETAILED DESCRIPTION:
This is a translational study. Patient will undergo standard treatment and tissue and blood samples will be taken at various time points:

Tissue: Fresh frozen (FF) and Formalin fixed paraffin embedded tissue (FFPE) will be collected at time of surgery/biopsy of a primary or a recurrent/metastatic tumour tissue.

Blood: Two types of study bloods (non-heparinised and Ethylenediaminetetraacetic acid (EDTA)) will be taken pre-neoadjuvant treatment (if applicable), pre- and post-operatively of primary and recurrent/ metastatic breast cancer (if recurrent/metastatic diagnosis and no biopsy/surgery required then study bloods will be taken prior to starting treatment).

Additional blood samples will be taken annually at follow-up visits for 5 years from primary cases and for up to 2 years from recurrent/metastatic cases.

Non-heparinised blood will be processed to serum. Clinical data will be collected at all times of biological sampling.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with primary breast cancer attending hospital for the resection of their tumour tissue

   Or

   -Patients with suspected or confirmed recurrent or metastatic breast cancer (Patient has a history of a biopsy- or surgically- (i.e. pathologically) confirmed primary breast cancer) attending hospital for the resection/biopsy and/or treatment of tumour tissue

   Or

   -Patient with suspected (but not necessarily biopsy confirmed) newly diagnosed stage 4 breast cancer attending hospital for the resection/biopsy and/or treatment of their tumour tissue
2. Patients receiving neoadjuvant treatment are also eligible (if applicable)
3. Patients have to be ≥ 18 years of age
4. Patients must be able to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All newly diagnosed breast cancer patients, recurrent and stage IV metastatic breast cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 1780 (Estimated)
Dates: Start 2013-02 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2038-01 (Estimated)

PRIMARY OUTCOMES:
Investigation of proteins and their pathways in primary breast cancer | 10 years
  Investigation of proteins and their pathways in primary breast cancer, which are associated with patient outcome.

SECONDARY OUTCOMES:
Comparison of the molecular profile between primary and recurrent/metastatic lesions in breast cancer | 10 years
Identification of novel molecular mechanisms of breast cancer recurrence | 10 years
  Identification of novel molecular mechanisms of breast cancer recurrence, therapy resistance and/or metastasis
Determination of novel potential molecular targets | 10 years
  Determination of novel potential molecular targets that can be used to develop future prevention and treatment advances in patients with breast cancer

CONTACTS AND LOCATIONS:
Locations (6):
- Ireland (6):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - St James's Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
  - University Hospital Limerick, Limerick
  - University Hospital Waterford, Waterford

REFERENCES:
- [Derived] Charmsaz S, Doherty B, Cocchiglia S, Vareslija D, Marino A, Cosgrove N, Marques R, Priedigkeit N, Purcell S, Bane F, Bolger J, Byrne C, O'Halloran PJ, Brett F, Sheehan K, Brennan K, Hopkins AM, Keelan S, Jagust P, Madden S, Martinelli C, Battaglini M, Oesterreich S, Lee AV, Ciofani G, Hill ADK, Young LS. ADAM22/LGI1 complex as a new actionable target for breast cancer brain metastasis. BMC Med. 2020 Nov 19;18(1):349. doi: 10.1186/s12916-020-01806-4. PMID 33208158
- [Derived] Charmsaz S, Hughes E, Bane FT, Tibbitts P, McIlroy M, Byrne C, Cocchiglia S, McBryan J, Hennessy BT, Dwyer RM, Kerin MJ, Hill AD, Young LS. S100beta as a serum marker in endocrine resistant breast cancer. BMC Med. 2017 Apr 12;15(1):79. doi: 10.1186/s12916-017-0836-2. PMID 28399921